CLINICAL TRIAL: NCT02344485
Title: Effect of Osteopathic Manipulative Medicine on Constipation in Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: New York Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BHS-1065
Record Dates: First submitted 2015-01-16; First posted 2015-01-26 (Estimated); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Parkinson's Disease; Constipation
MeSH Terms: conditions — Parkinson Disease; Constipation | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- OMM treatment (Experimental): Subject will receive osteopathic manipulative treatment protocol for constipation in Parkinson's disease once a week for 4 weeks, in addition to continuing with their routine care
  Interventions: Procedure: OMM treatment
- Control (No Intervention): Subjects will continue with their routine care. No OMM will be performed during this study period

INTERVENTIONS:
Procedure: OMM treatment — OMM is a gentle hands-on treatment that helps to reduce myofascial restrictions and improve joint range of motion. In doing so, it can address the mechanical, neurologic, and respiratory functions of the body
  Other Names: OMM (Osteopathic Manipulative Medicine); OMT (Osteopathic Manipulative Treatment); Osteopathic manipulation
  Arms: OMM treatment

SUMMARY:
The aim of this pilot study is to investigate the effect of Osteopathic Manipulative Medicine (OMM) in decreasing constipation symptoms in people with Parkinson's disease (PD). A second but optional aim is to determine if OMM changes the bacterial flora of the mouth and gut. OMM is a safe and gentle manual treatment provided by osteopathic physicians. All participants will receive OMM during the second half of the eleven week trial.

DETAILED DESCRIPTION:
PD is a progressive neurodegenerative disorder which includes motor and non-motor (autonomic) symptoms, such as constipation. OMM has been shown to improve constipation symptoms in non-diseased subjects and cerebral palsy subjects. Constipation will be measured before, during, and after treatment by a constipation scoring system (Cleveland Criteria) to measure the severity of constipation and by the Bristol Stool Scale to measure colonic transit time. The study subjects' assessment of their constipation symptoms (PAC-SYM) and quality of life (PAC-QOL) will also be measured throughout the study.

Studies have also shown that there is a difference in the gut and oral bacterial flora of constipated versus healthy adults, so subjects will be given the option to provide weekly stool samples for analysis to track bacterial colonies and to observe for any flora changes over the study period. This will provide data to determine if bacterial colonies in stool are altered by OMM.

The study will require ten weekly on-site visits over the course of eleven weeks. For the first half of the study, surveys and optional stool tests will be performed without OMM treatment for four weeks to obtain baseline data. For the second half of the study, all subjects will receive OMM for four weeks along with surveys and optional stool microbial tests to obtain the experimental data.

ELIGIBILITY:
Inclusion Criteria:

* Medically diagnosed with Parkinson's disease
* Medically diagnosed with constipation (according to Rome III criteria)
* Be over 40 years old

Exclusion Criteria:

* No diagnosis of Parkinson's disease
* No diagnosis of constipation that satisfies Rome III criteria
* Medically diagnosed with irritable bowel syndrome
* Another diagnosed cause for chronic constipation
* Currently pregnant
* Have another diagnosed neurologic condition (excluding headache or migraine, headache, migraine, dysautonomia, depression or other mood disorders (unless severe or uncontrolled), dementia or cognitive changes (unless severe), diffuse lewy body dementia, REM sleep behavior disorder, normal pressure hydrocephalus, multiple system atrophy P and C types, progressive supranuclear palsy, vascular parkinsonism, corticobasal ganglionic degeneration, and drug induced parkinsonism)
* Spinal cord abnormality or lesion
* Cancer of the gastrointestinal tract, abdomen, or pelvis
* Anemia that has not been evaluated
* Unexplained weight loss, fever, night sweats, rectal bleeding, or black stools in past 2 months
* Active hepatitis, infectious mononucleosis, or enlarged spleen
* Abdominal aortic aneurysm
* Congenital malformation of the gastrointestinal tract
* Abdominal or pelvic surgery within the past 6 weeks
* Unable or unwilling to receive OMT.
* Unable or unwilling to rate one's own stools using a visual chart or to bring a picture of one's stool to each visit

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-01-01; Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Constipation Scoring System (Cleveland Criteria) | 11 week period
  A standardized form measuring bowel movement patterns will be completed by the subject five times over the study period to see if there is a difference in constipation severity between the period with no OMT and the period with OMT

SECONDARY OUTCOMES:
Bristol Stool Scale | 11 week period
  A visual standardized stool chart will be used by the subject and study investigator nine times over the study period to visually categorize the shape of the stools to see if there is a difference in colonic transit time between the period with no OMT and the period with OMT
PAC-SYM© | 11 week period
  A standardized form will be completed by the subject five times over the study period to assess constipation symptoms to see if there is a difference between the period with no OMT and the period with OMT
PAC-QOL© | 11 week period
  A standardized form will be completed by the subject five times over the study period to assess the impact of constipation on daily life to see if there is a difference between the period with no OMT and the period with OMT

OTHER OUTCOMES:
Stool analysis | 11 week period
  Subjects will have the option of submitting stool samples up to five times over the study period to see if there is a difference in the gut bacterial flora between the period with no OMT and the period with OMT
Mouth analysis | 11 week period
  Subjects will have the option of submitting mouth samples (ie. cheek swabs) up to five times over the study period to see if there is a difference in the oral bacterial flora between the period with no OMT and the period with OMT

CONTACTS AND LOCATIONS:
Overall Officials: Jayme Mancini, D.O., Principal Investigator — New York Institute of Technology- Academic Health Care Center
Locations (1):
- New York Institute of Technology- Academic Health Care Center, Old Westbury, New York, United States

IPD SHARING:
Plan to Share IPD: No